CLINICAL TRIAL: NCT05251675
Title: Effect of Physician Peer Coaching on Burnout in Hospital-Based Physicians: A Pilot Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Prasanna Tadi, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-0144
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Burn Out
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching Group (Active Comparator): This arm will receive physician led coaching during the first 6 months of the study.
  Interventions: Behavioral: Physician Led Professional Coaching
- Non-Coached Group (Placebo Comparator): This arm will not receive physician led coaching until after the Coaching Group is finished with their coaching.
  Interventions: Behavioral: Delayed Physician Led Professional Coaching

INTERVENTIONS:
Behavioral: Physician Led Professional Coaching — This is a one-on-one intervention between a physician coach and an individual physician. This is meant to help coaches attain valued professional or personal development.
  Arms: Coaching Group
Behavioral: Delayed Physician Led Professional Coaching — This intervention will include professional one-on-one professional coaching delayed from the active comparator group.
  Arms: Non-Coached Group

SUMMARY:
The prevalence of burnout symptoms among physicians is high, especially for acute care physicians. Physician burn out is a long-term stress reaction marked by emotional exhaustion, depersonalization, and a lack of sense of personal accomplishment. The healthcare environment, due to its demanding pace and emotional intensity, puts physicians at high risk for burnout.

DETAILED DESCRIPTION:
Physician-Led Professional Coaching is a one-on-one intervention between a physician coach and an individual physician that is systematic, collaborative, future-focused, goal-oriented and is meant to help coaches attain valued professional or personal development. The trial will be conducted with 25 participants in an intervention cohort and 25 participants in a control. The intervention cohort will receive 6 individual coaching sessions over 6 months. Coaching sessions will use the CHEER acronym for conducting the coaching sessions: Celebrate, Hear, Executive coaching, Engage, and Recharge. The control group will be eligible for coaching sessions after the completing of the interventional arm. Physicians randomized to the control arm will be offered the same individualized coaching sessions as those that were in the intervention group. Te Maslach Burnout Inventory survey will be used to measure burnout and will be collected at baseline, 3 months, 6 months, and 9 months. The physician coach will be blinded to all survey data as it is being collected.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger Physician
* Practicing medicine at least 6 months in the Geisinger system

Exclusion Criteria:

* Currently seeking professional coaching sessions
* Planning to leave the Geisinger system within 1 year

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in burnout as measured by the Maslach Burnout Inventory | 9 months
  Providers will be asked to complete Maslach Burnout Inventory surveys at specific times during the coaching intervention. The surveys are based on a score of 0 (never) to 6 (every day) and used to determine if there is a reduction in provider burnout.

SECONDARY OUTCOMES:
Change in work environment factors contributing to burnout by Areas of Work life Survey | 9 months
  Providers will be asked to complete Areas of Work life surveys at specific times during the coaching intervention. The surveys are based on a score of 1 (Strongly Disagree) to 5 (Strongly Agree) and used to determine if there is a reduction in provider workload.

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Tadi, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Wilkes-Barre, Pennsylvania, United States